CLINICAL TRIAL: NCT06934967
Title: An Open-label, Single-arm, Multicenter, Phase 3 Study to Assess Pharmacokinetics, Safety and Tolerability of Iptacopan in Pediatric PNH Patients 2 to <18 Years of Age
Brief Title: Study to Assess the Pharmacokinetics, Safety, and Tolerability of Iptacopan in Pediatric PNH Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023I12201; 2024-515926-10 (EudraCT Number)
Record Dates: First submitted 2025-03-31; First posted 2025-04-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: Iptacopan,; PNH,; hemoglobin,; anemia
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Anemia | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LNP023-Cohort 1 (12 < 18 years old) (Experimental): Participants (12 to < 18 years old) will take iptacopan at the dose of 200 mg twice per day (in the morning and in the evening).
  Interventions: Drug: LNP023
- LNP023 -Cohort 2 (2 to < 12 years old) (Experimental): Participants (2 to < 12 years old) will be dosed based on weight at the Day 1 visit, initially. The study medication dose will be reassessed and re-adjusted as needed based on their weight at Week 12, 26, and 38.
  Interventions: Drug: LNP023

INTERVENTIONS:
Drug: LNP023 — Cohort 1-administered orally a dosing scheme of 200 mg twice-daily (two 100 mg capsules). Cohort 2- administered orally a dosing scheme based on weight at the Day 1, Week 12, 26 and 38.
  Other Names: Iptacopan

SUMMARY:
The purpose of this open-label, single arm, multicenter, phase 3 study is to assess the pharmacokinetics of iptacopan in pediatric patients and to assess whether iptacopan is safe and well tolerated when used for the treatment of pediatric paroxysmal nocturnal hemoglobinuria (PNH) patients 2 to < 18 years of age.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single arm study comprised of an up to a 8-week Screening Period, and a 26-week Treatment Period followed by a 26-week Extension Treatment Period.

This study will enroll a minimum of 12 pediatric patients 2 to < 18 years of age in a staggered manner into 3 cohorts: Cohort 1 (adolescents 12 to < 18 years of age, approximately 6 patients), Cohort 2a (6 to < 12 years of age, approximately 4 patients), and Cohort 2b (2 to < 6 years of age, approximately 2 patients).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 2 to < 18 years of age with a diagnosis of PNH confirmed by high-sensitivity flow cytometry with red blood cells (RBCs) and with white blood cells granulocytes/monocytes clone size ≥ 10%. The minimum body weight for patients in Cohort 1 is 35 kg.
* Patients being treated with anti-C5 therapy and who have been on a stable regimen (dose and interval) for at least 6 months prior to enrollment, may be screened and enrolled in the study and switched to iptacopan irrespective of their anemia and hemolysis status, at the discretion of the Principal Investigator.
* Patients who are anti-C5 treatment naive: mean hemoglobin level < 10 g/dL confirmed by central laboratory assessment during screening.
* Patients who are anti-C5 treatment naive: lactate dehydrogenase (LDH) > 1.5 × upper limit of normal (ULN) documented by at least 2 laboratory measurements 2 to 6 weeks apart during the screening period, one of which is to be done by the central lab.
* Vaccination against Neisseria meningitidis and Streptococcus pneumoniae infection is required prior to the start of study treatment. If the participant has not been previously vaccinated, or if a booster is required, vaccine should be given according to local guidelines at least 2 weeks prior to first study drug administration. If study treatment has to start earlier than 2 weeks post-vaccination, prophylactic antibiotic treatment should be initiated.
* Vaccination against Haemophilus influenzae is recommended, according to local guidelines, at least 2 weeks before iptacopan.

Exclusion Criteria:

* History of hypersensitivity to the study drug or its excipients or to drugs of similar chemical classes.
* Known or suspected hereditary complement deficiency at screening.
* History of hematopoietic stem cell transplantation (HSCT) or scheduled for HSCT within 52 weeks from enrollment into the study (Day 1).
* Patients with laboratory evidence of bone marrow failure (reticulocytes < 100 x 10 to the ninth/L; platelets < 30 × 10 to the ninth/L; neutrophils < 0.5 × 10 to the ninth/L).
* Active systemic bacterial, viral (including COVID-19), or fungal infection within 14 days prior to study drug administration.
* Presence of fever ≥ 38 °C (100.4 °F) within 7 days prior to study drug administration.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2031-11-19 (Estimated); Study Completion 2031-12-19 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 26 weeks
  Incidence and severity of AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.
PK parameter (Cmax) | Week 2
  Cmax is defined as the maximum (peak) observed concentration following a dose.
PK parameter (AUClast) | Week 2
  AUClast is the area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (tlast).
PK parameter (AUCtau) | Week 2
  AUCtau describes the area under the curve limited to the end of a dosing interval.
PK parameter (Ctrough) | Weeks 2, 4, 12 and 26
  Ctrough is the observed plasma concentration that is just prior to the beginning of, or at the end of a dosing interval.

SECONDARY OUTCOMES:
Change in hemoglobin (Hb) from baseline ≥1 g/dL (in the absence of RBC transfusions from Day 14). | Baseline, Week 26, Week 52
  To evaluate the proportion of patients who achieve an increase in hemoglobin levels from baseline of ≥ 1 g/dL at 26 weeks and at 52 weeks (in the absence of RBC transfusions from Day 14 until the end of the 26-week and 52-week treatment periods).
Change in Hb from baseline ≥2 g/dL (in the absence of RBC transfusions from Day 14). | Baseline, Week 26, Week 52
  To evaluate the proportion of patients who achieve an increase in hemoglobin levels from baseline of ≥ 2 g/dL at 26 weeks and at 52 weeks (in the absence of RBC transfusions from Day 14 until the end of the 26-week and 52-week treatment periods).
Normal Hb in the absence of red blood cell (RBC) transfusions from Day 14. | Week 26 and Week 52
  To evaluate the proportion of participants achieving hemoglobin normalization at 26 weeks and at 52 weeks (in the absence of RBC transfusions from Day 14 until the end of the 26-week and 52-week treatment periods).
Absence of packed-RBC transfusions and not meeting transfusion criteria from Day 14 at Week 26 and Week 52 | Week 26 and Week 52
  To evaluate transfusion avoidance as the proportion of participants who remain free from transfusions and do not meet transfusion criteria from Day 14 until the end of the 26-week treatment period and until the end of the 52-week treatment period.
Change from baseline in hemoglobin | Baseline, Week 26, Week 52
  To evaluate mean changes from baseline in hemoglobin at 26 weeks and at 52 weeks (evaluation of naive patients and prior anti-C5 treated patients, separately).
Change from baseline in lactate dehydrogenase (LDH) | Baseline, Week 26, Week 52
  To evaluate mean changes from baseline in LDH at 26 weeks and at 52 weeks (evaluation of naive patients and prior anti-C5 treated patients, separately).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (2):
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
- Brazil (5):
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Cali, Valle del Cauca Department, Colombia
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Genova, GE, Italy
- Novartis Investigative Site, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.